CLINICAL TRIAL: NCT05723575
Title: Behavioral and Neural Measures of Speech Motor Control
Brief Title: Modulation of Sensory Acuity With Transcranial Magnetic Stimulation (TMS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-1128 TMS (Exp 7); Protocol Version 8/25/2021 (Other: UW Madison); A481800 (Other: UW Madison); 1R01DC019134-01A1 (NIH)
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Results first posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Speech
Keywords: speech motor control; vocal learning
MeSH Terms: conditions — Speech | interventions — Transcranial Magnetic Stimulation; Electromyography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Adult Speakers (Experimental): healthy adult participants across the lifespan in three groups:18-35, 36-55, and 56+
  Interventions: Device: TMS; Behavioral: somatosensory acuity measurement

INTERVENTIONS:
Device: TMS — This paradigm uses theta-burst transcranial magnetic stimulation (tbTMS) to modulate the excitability of sensory cortices to examine the effect on sensory acuity and sensorimotor adaptation. Participants will complete three total sessions targeting primary somatosensory cortex (S1): one using intermittent theta-burst stimulation (iTBS), one using continuous theta-burst stimulation (cTBS), and one with sham stimulation.
  Other Names: transcranial magnetic stimulation (continuous and intermittent theta-burst stimulation), electromyography (EMG)
Behavioral: somatosensory acuity measurement — Somatosensory acuity will be measured through a tactile discrimination task using the corticalmetrics Brain Gauge. Participants lightly press their tongue onto two vibrating probes and report which one vibrated first or with greater amplitude.

SUMMARY:
The purpose of this research study is to understand how the brain processes and controls speech in healthy people. The investigators are doing this research because it will help identify the mechanisms that allow people to perceive their own speech errors and to learn new speech sounds, which may be applied to people who have communication disorders. 15 participants will be enrolled into this part of the study and can expect to be on study for 4 visits of 2-4 hours each.

DETAILED DESCRIPTION:
The overall study (Establishing the clinical utility of sensorimotor adaptation for speech rehabilitation) aims to understand how cognitive, perceptual, and motor processes are integrated in the control of speech movements. The investigators study how this complex skill is performed in healthy speakers to understand how this system functions, how this skill relates to the perception of speech, and what role different parts of the brain play in this process. Different studies look at how speech motor control is executed, maintained, and changed. Overall, the study will recruit 329 participants over the course of 5 years. Participants can expect to be on study for up to 3 weeks.

The entire study is composed of 8 experiments and 6 interventions. The present record represents the experiments involving transcranial magnetic stimulation (TMS), i.e. Experiment 7: Using TMS to alter somatosensory acuity.

This paradigm uses theta-burst transcranial magnetic stimulation (tbTMS) to modulate the excitability of sensory cortices to examine the effect on sensory acuity and sensorimotor adaptation. Participants will complete three total sessions targeting primary somatosensory cortex (S1): one using intermittent theta-burst stimulation (iTBS), one using continuous theta-burst stimulation (cTBS), and one with sham stimulation.

The effect of the stimulation on auditory acuity will be measured through a tactile discrimination task in which participants report the relative amplitude and/or timing of vibrating probes pressed lightly into the tongue using a custom device (a version of the Corticalmetrics Brain Gauge adapted to study the orofacial system).

ELIGIBILITY:
Inclusion Criteria (Control):

* English-speaking adults
* normal hearing and speech
* no history of stroke or neurological conditions

Exclusion Criteria:

* Native language other than English
* Any neurological disorders other than the disorder of interest
* Any history of hearing disorders
* Uncorrected vision problems that prevent participants from seeing visually-presented stimuli
* Significant cognitive impairments that prevent participants from carrying out the task or from giving informed consent
* Vulnerable populations (minors and prisoners)
* Additional exclusionary criteria for TMS:

  * Implanted paramagnetic materials (metal clips, plates, pacemakers, etc.)
  * Increased risk in the event of a seizure
  * Serious heart disease
  * Increased intracranial pressure
  * Pregnancy
  * History of seizures
  * Family history of epilepsy
  * Epileptogenic medications
  * Chronic or transient disruption of sleep (including jet lag)
  * History of fainting
  * Chronic or transient increase in stressful experiences
  * Use of illegal drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Niziolek, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Link to study record for experiment 5 [NCT05286658] — https://clinicaltrials.gov/study/NCT05286658

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 people provided data for this study from November 2022 to May 2023
Period: Overall Study
Arm/Group | Healthy Adult Speakers
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Adult Speakers
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 25 [18 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Somatosensory Acuity: Spatial Amplitude Discrimination Threshold (SDT)
Description: The investigators will measure thresholds in spatial amplitude discrimination (SDT). These thresholds represent the smallest difference that participants can detect in the amplitude of vibration on the tongue. Vibratory stimulation is delivered by the corticalmetrics Brain Gauge device, which has two probes, one on the left and one on the right side of the tongue. Participants will complete three total sessions targeting primary somatosensory cortex (S1): one using intermittent theta-burst stimulation (iTBS), one using continuous theta-burst stimulation (cTBS), and one with sham stimulation.
  Tactile acuity measured in this way is used as a proxy for full somatosensation, given the difficulty in measuring proprioception in the oral system. Tactile acuity has been suggested to be important for speech production, as tactile contact is maintained parasagittally during vowel production and tactile deprivation leads to imprecise speech movements.
Time Frame: up to 1 hour
Measure: Mean (Standard Error); unit: change in threshold (µm)
Arm/Group | Healthy Adult Speakers
Number analyzed (Participants) | 15
change in threshold (µm)
  SDT (cTBS) | 20.08 (7.37)
  SDT (iTBS) | -8.07 (3.74)
  SDT (sham) | 5.39 (5.59)
  SDT (control) | -2.81 (5.24)

2. Primary Outcome: Somatosensory Acuity: Temporal Discrimination Threshold (TDT)
Description: The investigators will measure thresholds in temporal discrimination (SDT). These thresholds represent the smallest difference that participants can detect in the timing of vibrations on the tongue. Vibratory stimulation is delivered by the corticalmetrics Brain Gauge device, which has two probes, one on the left and one on the right side of the tongue. Participants will complete three total sessions targeting primary somatosensory cortex (S1): one using intermittent theta-burst stimulation (iTBS), one using continuous theta-burst stimulation (cTBS), and one with sham stimulation.
  Tactile acuity measured in this way is used as a proxy for full somatosensation, given the difficulty in measuring proprioception in the oral system. Tactile acuity has been suggested to be important for speech production, as tactile contact is maintained parasagittally during vowel production and tactile deprivation leads to imprecise speech movements.
Time Frame: up to 1 hour
Measure: Mean (Standard Error); unit: change in threshold (ms)
Arm/Group | Healthy Adult Speakers
Number analyzed (Participants) | 15
change in threshold (ms)
  TDT (cTBS) | 0.41 (6.44)
  TDT (iTBS) | 5.80 (3.59)
  TDT (sham) | 4.54 (6.60)
  TDT (control) | -2.97 (6.25)

ADVERSE EVENTS:
Time Frame: Subjects participated in four sessions (each up to 4 hours) over the course of one month.
Description: Minimal risk basic science study, no adverse event collection plan required
Arm/Group | Healthy Adult Speakers
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT05723575/Prot_SAP_000.pdf